CLINICAL TRIAL: NCT00594867
Title: Does Acetaminophen Potentiate the Gastroduodenal Mucosal Injury of Aspirin? A Prospective, Randomized, Pilot Study.
Brief Title: The Effects of Aspirin and Acetaminophen on the Stomach in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Jay L. Goldstein, University of Illinois at Chicago
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-0459
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: Healthy; Volunteer
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Acetaminophen - 4 grams per day + Placebo
  Interventions: Drug: Acetaminophen - 4 grams per day + Placebo
- 2 (Active Comparator): Aspirin - 325 mg per day + Placebo
  Interventions: Drug: Aspirin - 325 mg per day + Placebo
- 3 (Experimental): Acetaminophen 4 gram per day + Aspirin 325 mg per day
  Interventions: Drug: Acetaminophen 4 gram per day + Aspirin 325 mg per day

INTERVENTIONS:
Drug: Acetaminophen - 4 grams per day + Placebo — Acetaminophen - 4 grams per day + Placebo
  Arms: 1
Drug: Aspirin - 325 mg per day + Placebo — Aspirin - 325 mg per day + Placebo
  Arms: 2
Drug: Acetaminophen 4 gram per day + Aspirin 325 mg per day — Acetaminophen 4 gram per day + Aspirin 325 mg per day
  Arms: 3

SUMMARY:
Aspirin is a medication commonly used to relieve minor pains. Aspirin has also been used to prevent heart attacks and strokes. Aspirin, however, can also cause damage to the stomach and/or intestinal lining leading to the development of erosions ("small sores") and/or ulcers ("large sores"). Erosions may cause bleeding ("bleeding ulcers") and/or perforations ("holes in the stomach"). Acetaminophen, often referred by the brand name, Tylenol, is also used to treat minor pains but is not commonly recognized to cause damage to the stomach lining.

Many patients often take both of these medications together. While the effects on the stomach lining of each medication, when used alone, are known, the effects of both medications, when used together, are not.

The purpose of this study is to show whether or not the collective effects of both aspirin and acetaminophen, when used together, increase the damage on the stomach lining when compared to either medication alone.

DETAILED DESCRIPTION:
Low dose aspirin is used for the primary and secondary prevention of cardiovascular thromboembolic events. As a non-selective inhibitor of cyclooxygenase, aspirin use results in irreversible COX-1 inhibition leading to impaired platelet aggregation. However, aspirin also inhibits COX-1 activity in the gastric mucosa by suppressing the synthesis of protective prostaglandins. In doing so, this creates a state of propensity for the development of aspirin-associated gastrointestinal ulcers and ulcer complications.

A high proportion of aspirin users also require concomitant use of anti-inflammatory medications for the treatment of pain and arthritis. However, evidence suggests that the risk of developing gastroduodenal ulcers and ulcer complications is significantly increased when aspirin is co-administered with other nonselective NSAIDs. In a previous study, concomitant aspirin (325 mg daily) in healthy subjects taking naproxen (500mg bid) was associated with endoscopic ulcer rates of 27.3% as compared to aspirin alone (7.6%). In a separate and independent trial of similar design, patients using 81 mg of aspirin in conjunction with daily naproxen also resulted in a higher incidence of gastric and duodenal ulcers than aspirin therapy alone. Beyond endoscopic ulcer rates, the risk of upper gastrointestinal hemorrhage has been reported to be substantially increased with concurrent administration of low-dose aspirin with nonselective NSAIDS. These data suggest that the gastrointestinal toxicity of combined aspirin with other NSAIDs may be more than additive.

ELIGIBILITY:
Inclusion Criteria:

1. Be a cooperative, healthy male or female between the ages of 18-75 inclusive.
2. Have a physical examination which reveals no clinically significant abnormalities at the screening visit.
3. Have fewer than 6 gastric or duodenal erosions visible on nasal endoscopy at Visit 2.
4. If the subject is female and of childbearing potential, she has been using effective contraception since the last date of her menses, will continue to use effective contraception during the study period, is not breast-feeding or lactating at screening and has had a negative urine pregnancy test at screening. Women who have been post-menopausal for less than 2 years will also require a urine pregnancy test at screening.
5. Have provided written informed consent prior for admission to this study.
6. H. pylori negative serologic exam prior to baseline nasal EGD.

Exclusion Criteria:

1. Active GI disease (e.g. IBD), or a history of GI ulcers or bleeding
2. History of gastric or intestinal surgery
3. Use of ASA, NSAIDs, coxibs, or acetaminophen at any dose within 2 weeks prior to the randomization visit of the study.
4. Positive FOBT at baseline.
5. Use of over-the-counter or prescription: sucralfate, antacids, H2-receptor antagonists, misoprostol, or proton pump inhibitors 4 weeks prior to enrollment and/or during the study
6. A known allergy to the topical anesthetic, lidocaine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence of combined gastric and duodenal ulcers, defined as >1 gastric, pyloric channel or duodenal ulcer (score 7), as determined by nasal upper GI endoscopy on day 7 of treatment. | 7 days

SECONDARY OUTCOMES:
Incidence of any gastric or duodenal ulcer (score 7) and any gastric and duodenal, gastric or duodenal erosions/ulcer (score 4-7) as determined by nasal upper endoscopy on day 7 of treatment. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jay L Goldstein, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] Patrono C, Garcia Rodriguez LA, Landolfi R, Baigent C. Low-dose aspirin for the prevention of atherothrombosis. N Engl J Med. 2005 Dec 1;353(22):2373-83. doi: 10.1056/NEJMra052717. No abstract available. PMID 16319386
- [Background] Weil J, Colin-Jones D, Langman M, Lawson D, Logan R, Murphy M, Rawlins M, Vessey M, Wainwright P. Prophylactic aspirin and risk of peptic ulcer bleeding. BMJ. 1995 Apr 1;310(6983):827-30. doi: 10.1136/bmj.310.6983.827. PMID 7711618
- [Background] Derry S, Loke YK. Risk of gastrointestinal haemorrhage with long term use of aspirin: meta-analysis. BMJ. 2000 Nov 11;321(7270):1183-7. doi: 10.1136/bmj.321.7270.1183. PMID 11073508
- [Background] Goldstein JL, Lowry SC, Lanza FL, Schwartz HI, Dodge WE. The impact of low-dose aspirin on endoscopic gastric and duodenal ulcer rates in users of a non-selective non-steroidal anti-inflammatory drug or a cyclo-oxygenase-2-selective inhibitor. Aliment Pharmacol Ther. 2006 May 15;23(10):1489-98. doi: 10.1111/j.1365-2036.2006.02912.x. PMID 16669964
- [Background] Sorensen HT, Mellemkjaer L, Blot WJ, Nielsen GL, Steffensen FH, McLaughlin JK, Olsen JH. Risk of upper gastrointestinal bleeding associated with use of low-dose aspirin. Am J Gastroenterol. 2000 Sep;95(9):2218-24. doi: 10.1111/j.1572-0241.2000.02248.x. PMID 11007221
- [Background] Cryer B, Feldman M. Cyclooxygenase-1 and cyclooxygenase-2 selectivity of widely used nonsteroidal anti-inflammatory drugs. Am J Med. 1998 May;104(5):413-21. doi: 10.1016/s0002-9343(98)00091-6. PMID 9626023
- [Background] Lanza FL, Codispoti JR, Nelson EB. An endoscopic comparison of gastroduodenal injury with over-the-counter doses of ketoprofen and acetaminophen. Am J Gastroenterol. 1998 Jul;93(7):1051-4. doi: 10.1111/j.1572-0241.1998.00327.x. PMID 9672328
- [Background] Jick H. Effects of aspirin and acetaminophen in gastrointestinal hemorrhage. Results from the Boston Collaborative Drug Surveillance Program. Arch Intern Med. 1981 Feb 23;141(3 Spec No):316-21. doi: 10.1001/archinte.141.3.316. PMID 6970559